CLINICAL TRIAL: NCT02648503
Title: Deep Neuromuscular Block and Sugammadex Versus Standard of Care on Quality of Recovery in Patient Undergo Elective Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Phan Ton Ngoc Vu, PhD. MD, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8616-138
Record Dates: First submitted 2015-12-07; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Neuromuscular Block
Keywords: Sugammadex; Post-operative Quality Recovery Scale (PQRS)
MeSH Terms: interventions — Rocuronium; Sugammadex; Atropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep neuromuscular block (Experimental): PTC=1-2
  Interventions: Drug: Deep neuromuscular block
- Moderate neuromuscular block (Active Comparator): TOF=1-2
  Interventions: Drug: Moderate neuromuscular block

INTERVENTIONS:
Drug: Deep neuromuscular block — Using rocuronium and reversal with sugammadex
  Other Names: Esmeron and Bridion
  Arms: Deep neuromuscular block
Drug: Moderate neuromuscular block — Using rocuronium and reversal with neostigmine (1 to 2 mg) and atropine (0.5 to 1 mg)
  Other Names: Esmeron and Neostigmin/Atropine
  Arms: Moderate neuromuscular block

SUMMARY:
Single center, prospective, randomized, single blinded, parallel group and controlled, assessor-blinded trial to compare the impact of Deep neuromuscular block and Sugammadex versus Standard of care on Quality of recovery in patient undergo elective laparoscopic cholecystectomy using PQRS at different time-point: 15 minutes (T15), 40 minutes (T40), one(D1) and three(D3) days after surgery

DETAILED DESCRIPTION:
* In the current study, the investigators investigate the effect of a deep NMB (TOF 0, PTC 1-2) with sugammadex against a moderate block (TOF 1-2) on quality of recovery in patient undergo elective laparoscopic cholecystectomy using PQRS at different time-point: 15 minutes (T15), 40 minutes (T40), one(D1) and three(D3) days after surgery.
* Based on a previous study comparing the Quality of recovery using PQRS between Neostigmine and Sugammadex, P. Amorim at al. showed that the percentage of patients fully awake at 40 min was 96.2% in the sugammadex group and 72.9% in the neostigmine group; the investigators expected the percentage of patient recovery at T40 will be 90% in group D (sugammadex) and 70% in group M (neostigmine)12. Recovery defined as return to the value of PQRS measured prior to surgery or higher. Using the formula for the sample size with α=0.05, Power: 80%, the sample size required per group is 60.
* Eligible patients will be randomly allocated into two groups using a computer-generated randomization before patients arrive to the operating room: Group D with deep, continuous neuromuscular blockade and Group M with moderate neuromuscular blockade.
* All information about group allocation, doses of rocuronium and sugammadex and neuromuscular data are recorded on a separate form and placed in a sealed opaque envelope when the patient is leaving the operating room. This will keep the personnel in the post-anesthesia care unit and the investigator collecting post-operative data blinded to group allocation.
* The investigators use acceleromyography (TOF-Watch SX) to monitor the level of neuromuscular blockage at the adductor pollicis muscle
* Involuntary movement will be recorded by anesthesia during surgery.
* Surgical condition will be rated by surgeons after surgery using five-point surgical condition scale (SRS)
* Hemodynamic changes using the noninvasive Nihon Konden (Nihon Konden, Japan), duration of surgery, drug dosages used during anesthesia, and duration from reversal to extubation, BIS, and ventilatory variables (tidal volume, respiratory rate, breathing pressure).
* Intra-abdominal pressure will be measured every 15 minutes from the peritoneal CO2 insufflation device. Pneumoperitoneum is obtained with insufflation of CO2 at 8 mmHg after the introduction of the trocars. In case of inadequate surgical conditions:

  * Increase of pre-set intra-abdominal pressure to 12-14 mmHg.
  * If still not adequate, patients will be given a bolus of rocuronium 0.075-0.15 mg/kg
  * If still not adequate, the surgeon will decide according to usual clinical practice.
* The intervention will be recorded by anesthesiologist and surgical condition rate will be measured at the time of surgery when they get worse.
* PQRS includes six domains of recovery: physiologic, nociceptive, emotive, activities of daily living, cognitive, and overall patient perspective. There is a series of questions in each domain2. PQRS data will be presented as percentage of patients that recovered for measurements taken at T15, T40, D1, and D3.
* Data of all patients that completed the baseline evaluation and T15 and T40 of the follow-up evaluations will be included in primary efficacy analysis.
* Continuous data will be presented as mean and standard deviation (SD) or median and range (minimum, maximum) and interquartile range (IQR, 25th 75th percentile). Categorical data will be presented as frequencies and percentages.
* The physiological domain data will be presented as mean and SD. The nociceptive domain data will be presented as mean with the 95% confidence intervals (CI).
* Categorical variables will be compared with the the Fisher exact test.
* For the comparison of continuous data, the Student's t test will be used. If there is substantial evidence of departures from normality, then the Mann-Whitney U-test will be performed as a sensitivity analysis.
* Data will be analyzed with the Statistical Package for the Social Sciences statistical software program. Statistical significance was set at P less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (> 18 years) scheduled for elective Laparoscopic Cholecystectomy with American Society of Anesthesiologist (ASA) class I-III in Hospital of University of Medicine and Pharmacy-Ho Chi Minh City

Exclusion Criteria:

* Patients with ASA class IV
* Age <18 years
* Inability to inform consent
* History or suspected with neuromuscular disorders
* Allergies to rocuronium or sugammadex, anesthetics or narcotics drugs
* A history of malignant hyperthermia
* A contraindication with neostigmine administration
* Pregnancy or breastfeeding
* Renal and liver insufficiency are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery | 40 minutes (T40) after the end of surgery
  The primary outcome is to access the differences of Quality of recovery in the overall recovery of the Post-operative Quality Recovery Scale (PQRS) instrument at 40 minutes (T40) after the end of surgery between Deep NMB (reversed with Sugammadex) and Standard of care in patients who undergo Laparoscopic Cholecystectomy.
  PQRS includes six domains of recovery: physiologic, nociceptive, emotive, activities of daily living, cognitive, and overall patient perspective. There is a series of questions in each domain. The Postoperative Quality Recovery Scale (PQRS) will be performed and recorded face-to-face by anesthesiologists in hospital and by telephone after discharge. The PQRS is completed prior to surgery to provide baseline values. Recovery is defined as returning to baseline values or better in each of the questions or assessments.

SECONDARY OUTCOMES:
Quality of recovery | 15 minutes (T15), and first day, 3 days after the end of surgery
  * The differences of Quality of recovery in the overall recovery of the PQRS instrument at 15 minutes (T15), and first day, 3 days after the end of surgery
  * The differences between each domain of PQRS instrument from 2 groups.
Shoulder tip pain | first hour, 6 hours and 24 hours after surgery
  using a 100 mm visual analogue scale (VAS) (0 indicating no pain and 100 worst imaginable pain)

OTHER OUTCOMES:
Surgical condition | intraoperation
  The satisfaction of surgeon with surgical condition from Deep Neuromuscular Block against Moderate Neuromuscular block. Surgeons will rate the surgical condition with a five-point surgical condition scale (SRS) ranging from 1= poor condition to 5= optimal surgical condition after the surgery
Time to discharge readiness | Every 20 min from the start of admission to the post-anesthesia care unit (PACU), up to 2 hours
  Time to discharge readiness from the post-anesthesia care unit (PACU) using Post Anesthesia Discharge Score System (PADSS)
Duration of operation | intraoperation
  Duration of surgery: from successful abdominal access with trocars to the skin closure Duration from reversal to extubation (TOF>0.9)

CONTACTS AND LOCATIONS:
Overall Officials: Vu TN Phan, PhD. MD, Principal Investigator — University medical center HCMC
Locations (1):
- Operation theathre, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes